CLINICAL TRIAL: NCT01928394
Title: A Phase 1/2, Open-label Study of Nivolumab Monotherapy or Nivolumab Combined With Ipilimumab in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: A Study of Nivolumab by Itself or Nivolumab Combined With Ipilimumab in Patients With Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-032; 2013-002844-10 (EudraCT Number)
Expanded Access: NCT02475382 (No longer available)
Record Dates: First submitted 2013-08-21; First posted 2013-08-23 (Estimated); Results first posted 2020-03-24 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Advanced or Metastatic Solid Tumors
MeSH Terms: interventions — Nivolumab; Ipilimumab; cobimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm N - Nivolumab (Experimental): Nivolumab 3 mg/kg solution intravenously every 2 weeks until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends
  Interventions: Biological: Nivolumab
- Arm N-I, Level 1: Nivolumab+Ipilimumab (Experimental): Nivolumab 1 mg/kg solution intravenously plus Ipilimumab 1 mg/kg solution every 3 weeks for 4 doses followed by Nivolumab 3 mg/kg every 2 weeks until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Arm N-I, Level 2: Nivolumab+Ipilimumab (Experimental): Nivolumab 1 mg/kg solution intravenously plus Ipilimumab 3 mg/kg every 3 weeks for 4 doses followed by nivolumab 3 mg/kg every 2 weeks until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Arm N-I, Level 2b: Nivolumab+Ipilimumab (Experimental): Nivolumab 3 mg/kg solution intravenously plus Ipilimumab 1 mg/kg every 3 weeks for 4 doses followed by nivolumab 3 mg/kg every 2 weeks until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Arm N-I, Level 2c: Nivolumab+Ipilimumab (Experimental): Nivolumab 3 mg/kg solution intravenously every 3 weeks combined with ipilimumab 1 mg/kg every 6 weeks until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Arm N-I, Level 2d: Nivolumab+Ipilimumab+Cobimetinib (Experimental): Nivolumab 3 mg/kg solution intravenously every 3 weeks combined with ipilimumab 1 mg/kg every 6 weeks and cobimetinib 60mg once daily 21days on/7 days off until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends
  Interventions: Biological: Nivolumab; Biological: Ipilimumab; Drug: Cobimetinib

INTERVENTIONS:
Biological: Nivolumab
  Other Names: BMS-936558; MDX-1106
Biological: Ipilimumab
  Other Names: Yervoy; BMS-734016; MDX-010
  Arms: Arm N-I, Level 1: Nivolumab+Ipilimumab; Arm N-I, Level 2: Nivolumab+Ipilimumab; Arm N-I, Level 2b: Nivolumab+Ipilimumab; Arm N-I, Level 2c: Nivolumab+Ipilimumab; Arm N-I, Level 2d: Nivolumab+Ipilimumab+Cobimetinib
Drug: Cobimetinib
  Other Names: Cotellic
  Arms: Arm N-I, Level 2d: Nivolumab+Ipilimumab+Cobimetinib

SUMMARY:
To investigate the safety and efficacy of nivolumab as a single agent or in combination with ipilimumab in 6 tumor types - triple-negative breast cancer (TNBC), gastric cancer (GC), pancreatic adenocarcinoma (PC), small cell lung cancer (SCLC), bladder cancer (BC), and ovarian cancer (OC). A combination of nivolumab with ipilimumab and cobimetinib is also investigated in PC.

DETAILED DESCRIPTION:
All tumor types are now closed for enrollment:

Triple Negative Breast Cancer

Gastric Cancer

Pancreatic Cancer

Small Cell Lung Cancer

Bladder Cancer

Ovarian Cancer

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Subjects with histologically or cytologically confirmed locally advanced or metastatic disease of the following tumor types:
* Triple Negative Breast Cancer
* Gastric Cancer
* Pancreatic Cancer
* Small Cell Lung Cancer
* Bladder Cancer
* Ovarian Cancer
* Subjects must have measurable disease
* Eastern Cooperative Oncology Group (ECOG) of 0 or 1
* Adequate hematological and organ function as confirmed by laboratory values

Exclusion Criteria:

* Active brain metastases or leptomeningeal metastases
* Subjects with active, known or suspected autoimmune disease
* Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of treatment
* Prior therapy with experimental anti-tumor vaccines; any T cell co-stimulation or checkpoint pathways, such as anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, including Ipilimumab; or other medicines specifically targeting T cell is also prohibited

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1163 (Actual)
Dates: Start 2013-10-24 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2024-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (38):
- United States (19):
  - Local Institution - 0047, Muscle Shoals, Alabama
  - Local Institution - 0044, Aurora, Colorado
  - Local Institution - 0015, New Haven, Connecticut
  - Local Institution - 0046, Gainesville, Florida
  - Local Institution - 0021, Tampa, Florida
  - Local Institution - 0001, Atlanta, Georgia
  - Local Institution - 0004, Baltimore, Maryland
  - Local Institution - 0005, Boston, Massachusetts
  - Local Institution - 0043, Boston, Massachusetts
  - Local Institution - 0049, Omaha, Nebraska
  - Local Institution - 0045, Mineola, New York
  - Local Institution - 0006, New York, New York
  - Local Institution - 0003, Charlotte, North Carolina
  - Local Institution - 0008, Durham, North Carolina
  - Local Institution - 0007, Portland, Oregon
  - Local Institution - 0011, Franklin, Tennessee
  - Local Institution - 0002, Nashville, Tennessee
  - Local Institution - 0009, Houston, Texas
  - Local Institution - 0042, Seattle, Washington
- Local Institution - 0038, Toronto, Ontario, Canada
- Local Institution - 0039, Copenhagen, Denmark
- Finland (2):
  - Local Institution - 0014, Helsinki, Uusimaa
  - Local Institution - 0036, Tampere
- Germany (4):
  - Local Institution - 0048, Bonn
  - Local Institution - 0026, Frankfurt
  - Local Institution - 0016, Heidelberg
  - Local Institution - 0050, Kassel
- Italy (4):
  - Local Institution - 0024, Bologna
  - Local Institution - 0019, Milan
  - Local Institution - 0020, Napoli
  - Local Institution - 0032, Padua
- Spain (4):
  - Local Institution - 0037, Barcelona
  - Local Institution - 0023, Madrid
  - Local Institution - 0017, Madrid
  - Local Institution - 0010, Madrid
- United Kingdom (3):
  - Local Institution - 0018, London, Greater London
  - Local Institution - 0012, Glasgow, Lanarkshire
  - Local Institution - 0013, Sutton, Surrey

REFERENCES:
- [Derived] Sharma P, Siefker-Radtke A, de Braud F, Basso U, Calvo E, Bono P, Morse MA, Ascierto PA, Lopez-Martin J, Brossart P, Rohrberg K, Mellado B, Fischer BS, Meadows-Shropshire S, Abdel Saci, Callahan MK, Rosenberg J. Nivolumab Alone and With Ipilimumab in Previously Treated Metastatic Urothelial Carcinoma: CheckMate 032 Nivolumab 1 mg/kg Plus Ipilimumab 3 mg/kg Expansion Cohort Results. J Clin Oncol. 2019 Jul 1;37(19):1608-1616. doi: 10.1200/JCO.19.00538. Epub 2019 May 17. PMID 31100038
- [Derived] Janjigian YY, Bendell J, Calvo E, Kim JW, Ascierto PA, Sharma P, Ott PA, Peltola K, Jaeger D, Evans J, de Braud F, Chau I, Harbison CT, Dorange C, Tschaika M, Le DT. CheckMate-032 Study: Efficacy and Safety of Nivolumab and Nivolumab Plus Ipilimumab in Patients With Metastatic Esophagogastric Cancer. J Clin Oncol. 2018 Oct 1;36(28):2836-2844. doi: 10.1200/JCO.2017.76.6212. Epub 2018 Aug 15. PMID 30110194
- [Derived] Teo MY, Seier K, Ostrovnaya I, Regazzi AM, Kania BE, Moran MM, Cipolla CK, Bluth MJ, Chaim J, Al-Ahmadie H, Snyder A, Carlo MI, Solit DB, Berger MF, Funt S, Wolchok JD, Iyer G, Bajorin DF, Callahan MK, Rosenberg JE. Alterations in DNA Damage Response and Repair Genes as Potential Marker of Clinical Benefit From PD-1/PD-L1 Blockade in Advanced Urothelial Cancers. J Clin Oncol. 2018 Jun 10;36(17):1685-1694. doi: 10.1200/JCO.2017.75.7740. Epub 2018 Feb 28. PMID 29489427
- [Derived] Sharma P, Callahan MK, Bono P, Kim J, Spiliopoulou P, Calvo E, Pillai RN, Ott PA, de Braud F, Morse M, Le DT, Jaeger D, Chan E, Harbison C, Lin CS, Tschaika M, Azrilevich A, Rosenberg JE. Nivolumab monotherapy in recurrent metastatic urothelial carcinoma (CheckMate 032): a multicentre, open-label, two-stage, multi-arm, phase 1/2 trial. Lancet Oncol. 2016 Nov;17(11):1590-1598. doi: 10.1016/S1470-2045(16)30496-X. Epub 2016 Oct 9. PMID 27733243
- [Derived] Antonia SJ, Lopez-Martin JA, Bendell J, Ott PA, Taylor M, Eder JP, Jager D, Pietanza MC, Le DT, de Braud F, Morse MA, Ascierto PA, Horn L, Amin A, Pillai RN, Evans J, Chau I, Bono P, Atmaca A, Sharma P, Harbison CT, Lin CS, Christensen O, Calvo E. Nivolumab alone and nivolumab plus ipilimumab in recurrent small-cell lung cancer (CheckMate 032): a multicentre, open-label, phase 1/2 trial. Lancet Oncol. 2016 Jul;17(7):883-895. doi: 10.1016/S1470-2045(16)30098-5. Epub 2016 Jun 4. PMID 27269741
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1131 participants were treated in total for TNBC, GC, PC, SCLC, BC and OC.
Groups:
- TNBC Arm N: Triple Negative Breast Cancer (TNBC) Nivolumab monotherapy (3 mg/kg) Q2W
- TNBC Arm N-I Dose Level 1: Triple Negative Breast Cancer (TNBC) Nivolumab (1 mg/kg) + ipilimumab (1 mg/kg) Q3W for 4 doses, then nivolumab (3 mg/kg) Q2W
- TNBC Arm N-I Dose Level 2: Triple Negative Breast Cancer (TNBC) Nivolumab (1 mg/kg) + ipilimumab (3 mg/kg) Q3W for 4 doses, then nivolumab (3 mg/kg) Q2W
- GC Arm N: Gastric Cancer (GC) Nivolumab 3 mg/kg Q2W
- GC Arm N-I Dose Level 1: Gastric Cancer(GC) Nivolumab (1 mg/kg) + ipilimumab (1 mg/kg) Q3W for 4 doses, then nivolumab (3 mg/kg) Q2W
- GC Arm N-I Dose Level 2: Gastric Cancer (GC) nivolumab (1 mg/kg) + ipilimumab (3 mg/kg) Q3W for 4 doses; then nivolumab 3 mg/kg Q2W
- GC Arm N-I Dose Level 2b: Gastric Cancer (GC) Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q3W for 4 doses, then Nivolumab (3 mg/kg) Q2W
- PC Arm N: Pancreatic cancer (PC) participants: Nivolumab 3 mg/kg Q2W
- PC Arm N-I Dose Level 1: Pancreatic cancer (PC) participants: Nivolumab 1 mg/kg + Ipilimumab 1 mg/kg Q3W for 4 doses, then Nivolumab (3 mg/kg) Q2W
- PC Arm N-I Dose Level 2: Pancreatic cancer (PC) participants: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Q3W for 4 doses, then Nivolumab (3 mg/kg) Q2W
- PC Arm N-I Dose Level 2d: Pancreatic cancer (PC) participants: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q6W for 4 doses + cobimetinib 60 mg po qd 21 days on/7 days off
- SCLC Arm N - Pre-expansion: Small cell lung cancer (SCLC) participants treated in Pre-expansion Cohort with Nivolumab 3 mg/kg Q2W
- SCLC Arm N-I Dose Level 2 - Pre-expansion: Small cell lung cancer (SCLC) treated participants in Pre-expansion cohort treated with Nivolumab (1 mg/kg) + ipilimumab (3 mg/kg) Q3W for 4 doses, then nivolumab (3 mg/kg) Q2W
- SCLC Arm N Expansion: Small cell lung cancer (SCLC) expansion cohort participants: Nivolumab monotherapy (3 mg/kg) Q2W
- SCLC Arm N-I Dose Level 2- Expansion: Small cell lung cancer (SCLC) expansion cohort participants Nivolumab (1 mg/kg) + ipilimumab (3 mg/kg) Q3W for 4 doses, then nivolumab (3 mg/kg) Q2W
- SCLC Arm N-I Dose Level 1 -: Small cell lung cancer (SCLC) participants treated with Nivolumab (1 mg/kg) + ipilimumab (1 mg/kg) Q3W for 4 doses, then nivolumab (3mg/kg) Q2W
- SCLC Arm N-I Dose Level 2b: Small cell lung cancer (SCLC) treated participants treated with Nivolumab (3 mg/kg) + ipilimumab (1 mg/kg) Q3W for 4 doses, then nivolumab (3 mg/kg) Q2W
- BC Arm N: Bladder cancer (BC) participants: Nivolumab 3 mg/kg Q2W
- BC Arm N-I Dose Level 2: Bladder cancer (BC) participants: Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg Q3W for 4 doses, then Nivolumab (3 mg/kg) Q2W
- BC Arm N-I Dose Level 2b: Bladder cancer (BC) participants: Nivolumab 3 mg/kg + Ipilimumab 1 mg/kg Q3W for 4 doses, then Nivolumab (3 mg/kg) Q2W
- OC Arm N-I Dose Level 2: Ovarian cancer (OC) participants:
  Nivolumab (1 mg/kg) + ipilimumab (3 mg/kg) Q3W for 4 doses, then nivolumab (3 mg/kg) Q2W
- OC Arm N-I Dose Level 2b: Ovarian cancer (OC) participants: Nivolumab (3 mg/kg) + ipilimumab (1 mg/kg) Q3W for 4 doses,then nivolumab (3 mg/kg) Q2W
- OC Arm N-I Dose Level 2c:: Ovarian cancer (OC) participants: Nivolumab (3 mg/kg) Q2W + ipilimumab (1 mg/kg) Q6W
Period: Treatment Period
Arm/Group | TNBC Arm N | TNBC Arm N-I Dose Level 1 | TNBC Arm N-I Dose Level 2 | GC Arm N | GC Arm N-I Dose Level 1 | GC Arm N-I Dose Level 2 | GC Arm N-I Dose Level 2b | PC Arm N | PC Arm N-I Dose Level 1 | PC Arm N-I Dose Level 2 | PC Arm N-I Dose Level 2d | SCLC Arm N - Pre-expansion | SCLC Arm N-I Dose Level 2 - Pre-expansion | SCLC Arm N Expansion | SCLC Arm N-I Dose Level 2- Expansion | SCLC Arm N-I Dose Level 1 - | SCLC Arm N-I Dose Level 2b | BC Arm N | BC Arm N-I Dose Level 2 | BC Arm N-I Dose Level 2b | OC Arm N-I Dose Level 2 | OC Arm N-I Dose Level 2b | OC Arm N-I Dose Level 2c:
Started (Started = Entering initial treatment or combination treatment after completion of monotherapy(MT)) | 18 | 3 | 18 | 59 | 3 | 49 | 52 | 18 | 3 | 18 | 30 | 98 | 61 | 147 | 96 | 3 | 55 | 78 | 92 | 104 | 41 | 43 | 42
Transition (Participants who will transition after completing MT due to disease progression (DP)) | 3 | 0 | 0 | 9 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 17 | 0 | 2 | 0 | 0 | 0 | 20 | 0 | 0 | 0 | 0 | 0
Transition- Continued (Participants who were transitioned to another treatment after disease progression (DP).) | 0 | 0 | 3 | 0 | 0 | 3 | 6 | 0 | 1 | 1 | 0 | 0 | 17 | 0 | 2 | 0 | 0 | 0 | 1 | 19 | 0 | 0 | 0
Completed (Completed = continuing treatment period) | 0 | 0 | 0 | 3 | 0 | 6 | 3 | 0 | 0 | 0 | 0 | 5 | 6 | 8 | 8 | 1 | 5 | 7 | 22 | 8 | 1 | 1 | 3
Not Completed | 18 | 3 | 18 | 56 | 3 | 43 | 49 | 18 | 3 | 18 | 30 | 93 | 55 | 139 | 88 | 2 | 50 | 71 | 70 | 96 | 40 | 42 | 39
Not completed — Disease progression | 17 | 2 | 12 | 48 | 3 | 25 | 38 | 16 | 3 | 11 | 22 | 73 | 38 | 118 | 59 | 1 | 43 | 56 | 50 | 71 | 30 | 31 | 31
Not completed — Study drug toxicity | 1 | 1 | 3 | 3 | 0 | 9 | 7 | 1 | 0 | 5 | 2 | 3 | 7 | 5 | 12 | 0 | 3 | 3 | 12 | 15 | 4 | 7 | 4
Not completed — AE unrelated to study drug | 0 | 0 | 2 | 3 | 0 | 5 | 1 | 0 | 0 | 2 | 0 | 12 | 6 | 13 | 6 | 1 | 1 | 6 | 3 | 5 | 1 | 1 | 0
Not completed — Participant request to stop therapy | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 0 | 3 | 2 | 1 | 2 | 4 | 0 | 1 | 3 | 1 | 1 | 3 | 1 | 3
Not completed — Participant withdrew consent | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 2 | 1 | 1 | 1 | 0 | 2 | 0
Not completed — Poor/non-compliance | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — other reason | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Not completed — Maximum clinical benefit | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Follow-up Period
Arm/Group | TNBC Arm N | TNBC Arm N-I Dose Level 1 | TNBC Arm N-I Dose Level 2 | GC Arm N | GC Arm N-I Dose Level 1 | GC Arm N-I Dose Level 2 | GC Arm N-I Dose Level 2b | PC Arm N | PC Arm N-I Dose Level 1 | PC Arm N-I Dose Level 2 | PC Arm N-I Dose Level 2d | SCLC Arm N - Pre-expansion | SCLC Arm N-I Dose Level 2 - Pre-expansion | SCLC Arm N Expansion | SCLC Arm N-I Dose Level 2- Expansion | SCLC Arm N-I Dose Level 1 - | SCLC Arm N-I Dose Level 2b | BC Arm N | BC Arm N-I Dose Level 2 | BC Arm N-I Dose Level 2b | OC Arm N-I Dose Level 2 | OC Arm N-I Dose Level 2b | OC Arm N-I Dose Level 2c:
Started (started = number of Participants regardless of continuing treatment or not.) | 15 | 3 | 18 | 50 | 3 | 49 | 52 | 16 | 3 | 18 | 30 | 81 | 61 | 145 | 96 | 3 | 55 | 58 | 92 | 104 | 41 | 43 | 42
Completed (completed = continuing to be followed) | 12 | 3 | 15 | 40 | 3 | 41 | 40 | 10 | 2 | 16 | 19 | 59 | 47 | 107 | 66 | 3 | 41 | 50 | 76 | 83 | 32 | 34 | 36
Not Completed | 3 | 0 | 3 | 10 | 0 | 8 | 12 | 6 | 1 | 2 | 11 | 22 | 14 | 38 | 30 | 0 | 14 | 8 | 16 | 21 | 9 | 9 | 6
Not completed — Participant withdrew consent | 3 | 0 | 1 | 4 | 0 | 2 | 5 | 1 | 0 | 0 | 5 | 8 | 2 | 12 | 7 | 0 | 5 | 3 | 2 | 7 | 4 | 6 | 2
Not completed — Death | 0 | 0 | 2 | 6 | 0 | 6 | 6 | 2 | 1 | 2 | 4 | 12 | 11 | 25 | 18 | 0 | 6 | 5 | 13 | 13 | 5 | 3 | 2
Not completed — other reason | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 2 | 1 | 0 | 1 | 4 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- SCLC Arm N Expansion: Small cell lung cancer (SCLC) expansion cohort participants:Nivolumab monotherapy (3 mg/kg) Q2W
- SCLC Arm N-I Dose Level 2- Expansion: Small cell lung cancer (SCLC) expansion cohort participants Nivolumab (1 mg/kg) + ipilimumab (3 mg/kg) Q3W for 4 doses, then nivolumab (3 mg/kg) Q2Wi
- OC Arm N-I Dose Level 2b:: Ovarian cancer (OC) participants: Nivolumab (3 mg/kg) + ipilimumab (1 mg/kg) Q3W for 4 doses,then nivolumab (3 mg/kg) Q2W
- Total: Total of all reporting groups
Arm/Group | TNBC Arm N | TNBC Arm N-I Dose Level 1 | TNBC Arm N-I Dose Level 2 | GC Arm N | GC Arm N-I Dose Level 1 | GC Arm N-I Dose Level 2 | GC Arm N-I Dose Level 2b | PC Arm N | PC Arm N-I Dose Level 1 | PC Arm N-I Dose Level 2 | PC Arm N-I Dose Level 2d | SCLC Arm N - Pre-expansion | SCLC Arm N-I Dose Level 2 - Pre-expansion | SCLC Arm N Expansion | SCLC Arm N-I Dose Level 2- Expansion | SCLC Arm N-I Dose Level 1 - | SCLC Arm N-I Dose Level 2b | BC Arm N | BC Arm N-I Dose Level 2 | BC Arm N-I Dose Level 2b | OC Arm N-I Dose Level 2 | OC Arm N-I Dose Level 2b: | OC Arm N-I Dose Level 2c: | Total
Number analyzed (Participants) | 18 | 3 | 18 | 59 | 3 | 49 | 52 | 18 | 3 | 18 | 30 | 98 | 61 | 147 | 96 | 3 | 55 | 78 | 92 | 104 | 41 | 43 | 42 | 1131
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: All Treated Participants
  Years | 53.3 (11.9) | 52.7 (9.5) | 49.1 (9.0) | 57.2 (10.99) | 67.0 (9.54) | 53.2 (12.58) | 56.4 (13.40) | 63.2 (9.70) | 58.3 (9.87) | 64.1 (9.21) | 62.1 (11.51) | 62.6 (8.50) | 63.9 (9.94) | 62.8 (9.09) | 63.7 (9.06) | 59.3 (6.7) | 60.1 (7.74) | 64.1 (10.86) | 63.9 (9.54) | 64.1 (9.69) | 56.7 (11.1) | 59.6 (10.9) | 58.7 (12.2) | 61.2 (10.7)
Age, Customized [Number; unit: Participants] — Age categorization Population: All Treated Participants
  Participants
    < 65 | 16 | 3 | 18 | 42 | 1 | 39 | 35 | 5 | 2 | 9 | 13 | 55 | 27 | 82 | 47 | 2 | 38 | 37 | 47 | 57 | 30 | 26 | 25 | 656
    >= 65 and < 75 | 1 | 0 | 0 | 15 | 1 | 8 | 12 | 12 | 1 | 7 | 14 | 34 | 27 | 51 | 39 | 1 | 17 | 31 | 34 | 29 | 10 | 14 | 12 | 370
    >= 75 | 1 | 0 | 0 | 2 | 1 | 2 | 5 | 1 | 0 | 2 | 3 | 9 | 7 | 14 | 10 | 0 | 0 | 10 | 11 | 18 | 1 | 3 | 5 | 105
    >= 65 | 2 | 0 | 0 | 17 | 2 | 10 | 17 | 13 | 1 | 9 | 17 | 43 | 34 | 65 | 49 | 1 | 17 | 41 | 45 | 47 | 11 | 17 | 17 | 475
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All treated Participants
  Participants
    Female | 18 | 3 | 18 | 14 | 1 | 15 | 7 | 5 | 2 | 8 | 12 | 37 | 26 | 61 | 35 | 1 | 23 | 24 | 18 | 23 | 41 | 43 | 42 | 477
    Male | 0 | 0 | 0 | 45 | 2 | 34 | 45 | 13 | 1 | 10 | 18 | 61 | 35 | 86 | 61 | 2 | 32 | 54 | 74 | 81 | 0 | 0 | 0 | 654
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: All Treated Participants
  Participants
    Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 4 | 1 | 1 | 1 | 18
    Not Hispanic or Latino | 10 | 3 | 9 | 41 | 2 | 29 | 35 | 16 | 3 | 13 | 28 | 63 | 47 | 97 | 55 | 2 | 26 | 59 | 38 | 73 | 26 | 29 | 32 | 736
    Unknown or Not Reported | 8 | 0 | 9 | 17 | 1 | 19 | 15 | 2 | 0 | 4 | 2 | 32 | 14 | 50 | 41 | 1 | 28 | 17 | 54 | 27 | 14 | 13 | 9 | 377
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All Treated Participnats
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Asian | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 4 | 2 | 0 | 1 | 18
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 3 | 0 | 1 | 3 | 0 | 1 | 1 | 1 | 0 | 1 | 4 | 3 | 1 | 7 | 5 | 1 | 0 | 4 | 3 | 4 | 1 | 0 | 2 | 46
    White | 14 | 3 | 17 | 56 | 3 | 46 | 50 | 16 | 3 | 16 | 23 | 91 | 60 | 134 | 87 | 2 | 54 | 72 | 87 | 90 | 37 | 43 | 38 | 1042
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 4 | 3 | 0 | 1 | 1 | 1 | 6 | 1 | 0 | 1 | 24

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate ( ORR )
Description: The number of participants with a best overall response (BOR) of complete response (CR) or partial response (PR) divided by the number of treated participants.
Time Frame: 60 months
Population: All Treated Participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- SCLC Arm N- All Treated: Small cell lung cancer (SCLC) for all treated participants with Nivolumab 3 mg/kg Q2W
- SCLC Arm N-I Dose Level 2 - All Treated: Small cell lung cancer (SCLC) all treated participants with Nivolumab (1 mg/kg) + ipilimumab (3 mg/kg) Q3W for 4 doses
Arm/Group | TNBC Arm N | TNBC Arm N-I Dose Level 1 | TNBC Arm N-I Dose Level 2 | GC Arm N | GC Arm N-I Dose Level 1 | GC Arm N-I Dose Level 2 | GC Arm N-I Dose Level 2b | PC Arm N | PC Arm N-I Dose Level 1 | PC Arm N-I Dose Level 2 | PC Arm N-I Dose Level 2d | SCLC Arm N - Pre-expansion | SCLC Arm N-I Dose Level 2 - Pre-expansion | SCLC Arm N Expansion | SCLC Arm N-I Dose Level 2- Expansion | SCLC Arm N-I Dose Level 1 - | SCLC Arm N-I Dose Level 2b | SCLC Arm N- All Treated | SCLC Arm N-I Dose Level 2 - All Treated | BC Arm N | BC Arm N-I Dose Level 2 | BC Arm N-I Dose Level 2b | OC Arm N-I Dose Level 2 | OC Arm N-I Dose Level 2b: | OC Arm N-I Dose Level 2c:
Number analyzed (Participants) | 18 | 3 | 18 | 59 | 3 | 49 | 52 | 18 | 3 | 18 | 30 | 98 | 61 | 147 | 96 | 3 | 55 | 245 | 157 | 78 | 92 | 104 | 41 | 43 | 42
Percentage of Participants | 5.6 [0.1 to 27.3] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 18.5] | 11.9 [4.9 to 22.9] | 0.0 [0.0 to 70.8] | 24.5 [13.3 to 38.9] | 7.7 [2.1 to 18.5] | 0.0 [0 to 18.5] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 18.5] | 6.7 [0.8 to 22.1] | 13.3 [7.3 to 21.6] | 26.2 [15.8 to 39.1] | 11.6 [6.9 to 17.9] | 21.9 [14.1 to 31.5] | 33.3 [0.8 to 90.6] | 18.2 [9.1 to 30.9] | 11.8 [8.1 to 16.6] | 22.3 [16.0 to 29.6] | 25.6 [16.4 to 36.8] | 38.0 [28.1 to 48.8] | 26.9 [18.7 to 36.5] | 12.2 [4.1 to 26.2] | 7.0 [1.5 to 19.1] | 9.5 [2.7 to 22.6]
Statistical Analysis 1: Comparison: SCLC Arm N Expansion vs SCLC Arm N-I Dose Level 2- Expansion; SCLC Arm N Expansion as compare to SCLC Arm N-I Dose Level 2- Expansion; Test type: Superiority; p = 0.0309, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.12, 95% CI 2-sided [1.06 to 4.26]

ADVERSE EVENTS:
Time Frame: Includes events reported between first dose and 30 days (AEs) or 100 days (SAEs) after last dose of study therapy
Groups:
- SCLC Arm N: Small cell lung cancer (SCLC) pre-expansion and expansion cohort participants: Nivolumab monotherapy (3 mg/kg) Q2W
- SCLC Arm N-I Dose Level 2: Small cell lung cancer (SCLC) pre-expansion and expansion cohort participants: Nivolumab (1 mg/kg) + ipilimumab (3 mg/kg) Q3W for 4 doses, then nivolumab (3 mg/kg) Q2Wi
- SCLC Arm N-I Dose Level 1: Small cell lung cancer (SCLC) participants treated with Nivolumab (1 mg/kg) + ipilimumab (1 mg/kg) Q3W for 4 doses, then nivolumab (3mg/kg) Q2W
- OC Arm N-I Dose Level 2c: Ovarian cancer (OC) participants: Nivolumab (3 mg/kg) Q2W + ipilimumab (1 mg/kg) Q6W
Arm/Group | TNBC Arm N | TNBC Arm N-I Dose Level 1 | TNBC Arm N-I Dose Level 2 | GC Arm N | GC Arm N-I Dose Level 1 | GC Arm N-I Dose Level 2 | GC Arm N-I Dose Level 2b | PC Arm N | PC Arm N-I Dose Level 1 | PC Arm N-I Dose Level 2 | PC Arm N-I Dose Level 2d | SCLC Arm N | SCLC Arm N-I Dose Level 2 | SCLC Arm N-I Dose Level 1 | SCLC Arm N-I Dose Level 2b | BC Arm N | BC Arm N-I Dose Level 2 | BC Arm N-I Dose Level 2b | OC Arm N-I Dose Level 2 | OC Arm N-I Dose Level 2b | OC Arm N-I Dose Level 2c
All-Cause Mortality (participants affected / at risk) | 17/18 | 3/3 | 18/18 | 53/59 | 3/3 | 42/49 | 50/52 | 18/18 | 3/3 | 18/18 | 24/30 | 212/245 | 136/157 | 3/3 | 45/55 | 60/78 | 54/92 | 82/104 | 33/41 | 37/43 | 34/42
Serious Adverse Events (participants affected / at risk) | 9/18 | 2/3 | 11/18 | 32/59 | 1/3 | 37/49 | 34/52 | 10/18 | 3/3 | 11/18 | 16/30 | 129/245 | 111/157 | 2/3 | 32/55 | 41/78 | 62/92 | 72/104 | 24/41 | 31/43 | 29/42
Other Adverse Events (participants affected / at risk) | 18/18 | 3/3 | 17/18 | 58/59 | 3/3 | 47/49 | 49/52 | 18/18 | 3/3 | 17/18 | 29/30 | 226/245 | 147/157 | 3/3 | 53/55 | 77/78 | 85/92 | 100/104 | 38/41 | 40/43 | 41/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TNBC Arm N (N=18) | TNBC Arm N-I Dose Level 1 (N=3) | TNBC Arm N-I Dose Level 2 (N=18) | GC Arm N (N=59) | GC Arm N-I Dose Level 1 (N=3) | GC Arm N-I Dose Level 2 (N=49) | GC Arm N-I Dose Level 2b (N=52) | PC Arm N (N=18) | PC Arm N-I Dose Level 1 (N=3) | PC Arm N-I Dose Level 2 (N=18) | PC Arm N-I Dose Level 2d (N=30) | SCLC Arm N (N=245) | SCLC Arm N-I Dose Level 2 (N=157) | SCLC Arm N-I Dose Level 1 (N=3) | SCLC Arm N-I Dose Level 2b (N=55) | BC Arm N (N=78) | BC Arm N-I Dose Level 2 (N=92) | BC Arm N-I Dose Level 2b (N=104) | OC Arm N-I Dose Level 2 (N=41) | OC Arm N-I Dose Level 2b (N=43) | OC Arm N-I Dose Level 2c (N=42)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pericardial haemorrhage (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 2 | 1 | 1
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypopituitarism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Endocrine ophthalmopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 3 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 3 | 3 | 3 | 2 | 3 | 4
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 3
Autoimmune colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 1 | 0 | 2 | 0 | 0 | 6 | 0 | 1 | 2 | 3 | 4 | 1 | 1 | 1
Colonic fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 5 | 0 | 1 | 0 | 1 | 1 | 3 | 7 | 0 | 1 | 4 | 10 | 7 | 2 | 3 | 2
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 2 | 3 | 4
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 0 | 0 | 2 | 4 | 1 | 0 | 0 | 1 | 1 | 4 | 2 | 3 | 2
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 2 | 5 | 1 | 3 | 3
Adverse event (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Cyst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 2 | 0 | 3 | 3 | 2 | 0 | 1 | 3 | 4 | 2 | 0 | 0 | 2 | 4 | 7 | 0 | 1 | 1
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Steatohepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspergillus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Biliary sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Meningitis aseptic (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peritoneal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 13 | 7 | 0 | 3 | 1 | 2 | 0 | 0 | 2 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Salmonellosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Systemic candida (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 3 | 5 | 3 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral diarrhoea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaesthetic complication neurological (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Radiation injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 4 | 2 | 1 | 0 | 1 | 0 | 3 | 2 | 0 | 0 | 0 | 2 | 6 | 1 | 2 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 2 | 5 | 1 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 3 | 6 | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Type 3 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 2 | 9 | 1 | 7 | 7 | 3 | 2 | 4 | 3 | 54 | 35 | 1 | 13 | 7 | 13 | 10 | 2 | 2 | 4
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Limbic encephalitis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myasthenic syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraparesis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device leakage (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 5 | 4 | 3 | 0 | 1 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 0
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prerenal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urethral obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 5 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 6 | 3 | 0 | 0 | 3 | 2 | 8 | 0 | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 5 | 1 | 0 | 1 | 1 | 0 | 0 | 4 | 0 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 0 | 1 | 4 | 0 | 0 | 0 | 1 | 6 | 7 | 0 | 1 | 1 | 4 | 3 | 0 | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Poor venous access (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TNBC Arm N (N=18) | TNBC Arm N-I Dose Level 1 (N=3) | TNBC Arm N-I Dose Level 2 (N=18) | GC Arm N (N=59) | GC Arm N-I Dose Level 1 (N=3) | GC Arm N-I Dose Level 2 (N=49) | GC Arm N-I Dose Level 2b (N=52) | PC Arm N (N=18) | PC Arm N-I Dose Level 1 (N=3) | PC Arm N-I Dose Level 2 (N=18) | PC Arm N-I Dose Level 2d (N=30) | SCLC Arm N (N=245) | SCLC Arm N-I Dose Level 2 (N=157) | SCLC Arm N-I Dose Level 1 (N=3) | SCLC Arm N-I Dose Level 2b (N=55) | BC Arm N (N=78) | BC Arm N-I Dose Level 2 (N=92) | BC Arm N-I Dose Level 2b (N=104) | OC Arm N-I Dose Level 2 (N=41) | OC Arm N-I Dose Level 2b (N=43) | OC Arm N-I Dose Level 2c (N=42)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 4 | 19 | 1 | 12 | 17 | 5 | 1 | 8 | 3 | 37 | 26 | 0 | 10 | 27 | 18 | 30 | 4 | 10 | 8
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 1 | 1 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 5 | 3 | 0 | 6 | 3 | 0 | 1 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 2 | 1 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 6 | 1 | 0 | 1 | 3 | 2 | 2 | 3 | 1 | 3
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 4 | 5 | 0 | 2 | 0 | 3 | 1 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 3
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 5 | 2 | 0 | 2 | 1 | 0 | 2 | 0 | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 1 | 0 | 2 | 2 | 1 | 2 | 5
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1
Hyperthyroidism (Endocrine disorders) | 2 | 0 | 0 | 5 | 0 | 4 | 4 | 0 | 0 | 2 | 1 | 7 | 22 | 0 | 5 | 4 | 9 | 13 | 6 | 3 | 3
Hypogonadism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 1 | 3 | 0 | 6 | 4 | 2 | 0 | 0 | 2 | 14 | 24 | 0 | 6 | 9 | 14 | 16 | 7 | 10 | 8
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thyroid disorder (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 1 | 3 | 0 | 3 | 3 | 1 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dry eye (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 3 | 0 | 3 | 2 | 2 | 0 | 0
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 2 | 1 | 0 | 0 | 1
Photopsia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 1 | 2 | 6 | 6 | 1 | 1 | 3 | 6 | 1 | 1 | 2 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 6 | 1 | 3 | 5 | 2 | 0 | 2 | 1 | 8 | 7 | 0 | 1 | 1 | 2 | 5 | 3 | 2 | 7
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 3 | 17 | 0 | 7 | 9 | 5 | 1 | 5 | 5 | 17 | 19 | 1 | 6 | 14 | 15 | 21 | 17 | 19 | 11
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 7 | 0 | 5 | 6 | 0 | 0 | 2 | 1 | 9 | 7 | 0 | 3 | 5 | 3 | 6 | 3 | 3 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 8 | 1 | 4 | 7 | 2 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 4 | 7 | 6
Colitis (Gastrointestinal disorders) | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 9 | 1 | 1 | 1 | 3 | 3 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 5 | 15 | 2 | 9 | 16 | 6 | 0 | 6 | 5 | 49 | 34 | 0 | 12 | 16 | 19 | 28 | 9 | 14 | 10
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 11 | 17 | 1 | 15 | 8 | 4 | 1 | 10 | 21 | 54 | 45 | 2 | 17 | 17 | 44 | 38 | 13 | 19 | 16
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0 | 3 | 7 | 0 | 1 | 2 | 0 | 12 | 5 | 0 | 5 | 8 | 11 | 13 | 5 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 2 | 0 | 1 | 0 | 0 | 2 | 3 | 8 | 3 | 1 | 1 | 2 | 5 | 4 | 3 | 2 | 4
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 9 | 0 | 1 | 13 | 0 | 1 | 0 | 1 | 8 | 8 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 0 | 1 | 2 | 1 | 0 | 1 | 3 | 2 | 6 | 0 | 0 | 3 | 0 | 2 | 0 | 1 | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 4 | 1 | 0 | 1 | 1 | 6 | 5 | 0 | 1 | 1 | 1 | 4 | 1 | 0 | 4
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 1 | 6 | 21 | 3 | 15 | 14 | 6 | 0 | 10 | 12 | 55 | 38 | 2 | 17 | 23 | 25 | 33 | 16 | 21 | 18
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Steatorrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 9 | 4 | 0 | 1 | 4 | 7 | 9 | 4 | 1 | 3
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 3 | 1 | 1 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 5 | 18 | 2 | 9 | 16 | 7 | 1 | 4 | 15 | 37 | 26 | 0 | 11 | 13 | 19 | 19 | 9 | 13 | 11
Asthenia (General disorders) | 0 | 1 | 1 | 4 | 0 | 5 | 7 | 0 | 0 | 0 | 3 | 28 | 19 | 0 | 12 | 4 | 5 | 6 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 13 | 4 | 0 | 4 | 2 | 2 | 1 | 0 | 0 | 0
Chills (General disorders) | 2 | 0 | 0 | 5 | 0 | 2 | 2 | 3 | 0 | 5 | 5 | 8 | 8 | 0 | 3 | 4 | 11 | 1 | 3 | 3 | 4
Early satiety (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Face oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 8 | 2 | 7 | 32 | 2 | 22 | 28 | 11 | 1 | 13 | 22 | 89 | 67 | 2 | 25 | 46 | 36 | 52 | 21 | 24 | 27
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 9 | 5 | 1 | 2 | 1 | 1 | 3 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperpyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 1 | 1 | 1 | 2 | 7 | 0 | 1 | 1
Localised oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 2 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 1 | 1 | 2 | 0 | 3 | 6 | 0 | 1 | 2 | 3 | 3 | 3 | 0 | 2
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 2 | 2 | 3 | 0 | 0 | 0 | 1 | 4 | 2 | 1 | 2
Nodule (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 11 | 6 | 0 | 1 | 1 | 1 | 4 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 3 | 7 | 0 | 5 | 6 | 5 | 1 | 3 | 9 | 18 | 19 | 0 | 3 | 13 | 18 | 22 | 7 | 8 | 5
Pain (General disorders) | 1 | 0 | 0 | 4 | 0 | 3 | 6 | 1 | 0 | 1 | 1 | 8 | 10 | 0 | 0 | 6 | 12 | 12 | 3 | 2 | 3
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 4 | 0 | 4 | 16 | 0 | 10 | 14 | 5 | 0 | 6 | 12 | 14 | 20 | 0 | 5 | 11 | 29 | 17 | 9 | 9 | 7
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tenderness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 3
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacterial disease carrier (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 0 | 0 | 6 | 1 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 1
Helicobacter gastritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 1 | 0 | 2 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 5 | 2 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 7 | 7 | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 6 | 4 | 0 | 1 | 3 | 1 | 2 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 4 | 0 | 0 | 5 | 0 | 0 | 0 | 1 | 6 | 6 | 0 | 2 | 0 | 2 | 2 | 0 | 2 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 6 | 2 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 4 | 4 | 1 | 1 | 4 | 2 | 3 | 1 | 1 | 2
Skin infection (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 2 | 2 | 2 | 0 | 0 | 2 | 12 | 7 | 0 | 4 | 9 | 2 | 6 | 0 | 2 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 3 | 0 | 1 | 1 | 0 | 0 | 1 | 3 | 12 | 14 | 1 | 1 | 8 | 10 | 12 | 3 | 1 | 8
Accidental device ingestion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 6 | 5 | 0 | 0 | 1 | 2 | 3 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 11 | 7 | 1 | 4 | 3 | 2 | 3 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 14 | 1 | 0 | 2 | 3 | 0 | 1 | 3 | 2 | 3
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Activated partial thromboplastin time (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1 | 7 | 6 | 0 | 11 | 5 | 3 | 0 | 5 | 2 | 26 | 20 | 0 | 4 | 8 | 15 | 20 | 9 | 4 | 9
Amylase increased (Investigations) | 0 | 0 | 2 | 3 | 0 | 3 | 2 | 0 | 0 | 2 | 1 | 14 | 18 | 0 | 3 | 7 | 9 | 15 | 3 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 7 | 8 | 0 | 9 | 4 | 5 | 1 | 5 | 3 | 27 | 25 | 0 | 4 | 6 | 11 | 19 | 8 | 6 | 10
Blood alkaline phosphatase increased (Investigations) | 2 | 1 | 3 | 6 | 0 | 7 | 4 | 3 | 1 | 7 | 5 | 15 | 13 | 0 | 3 | 7 | 2 | 15 | 3 | 3 | 4
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 2 | 0 | 2 | 2 | 3 | 0 | 3 | 2 | 9 | 8 | 0 | 0 | 1 | 0 | 7 | 0 | 0 | 3
Blood calcium decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 1 | 1 | 0 | 2 | 2 | 1 | 0 | 1 | 1 | 9 | 10 | 0 | 1 | 16 | 8 | 16 | 2 | 3 | 3
Blood lactic acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 3 | 5 | 0 | 1 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 4 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 2 | 2 | 0 | 7 | 4 | 1 | 0 | 4 | 0 | 21 | 15 | 0 | 2 | 14 | 9 | 15 | 4 | 4 | 4
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 5 | 3 | 9 | 2 | 0 | 2
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 3 | 0 | 6 | 2 | 0 | 0 | 6 | 1 | 11 | 0 | 1 | 1
Transaminases increased (Investigations) | 1 | 0 | 1 | 2 | 0 | 3 | 1 | 0 | 0 | 2 | 0 | 3 | 1 | 0 | 2 | 1 | 2 | 3 | 0 | 0 | 3
Troponin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 2 | 0 | 3 | 8 | 0 | 3 | 8 | 1 | 1 | 4 | 1 | 15 | 24 | 0 | 7 | 5 | 23 | 16 | 6 | 4 | 5
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 4 | 4 | 0 | 0 | 1 | 4 | 4 | 1 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 4 | 2 | 4 | 0 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0 | 2 | 21 | 2 | 14 | 19 | 6 | 0 | 7 | 11 | 67 | 50 | 1 | 15 | 14 | 21 | 36 | 10 | 11 | 13
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 9 | 0 | 3 | 4 | 4 | 1 | 2 | 2 | 14 | 15 | 0 | 5 | 4 | 2 | 6 | 2 | 5 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 3 | 0 | 8 | 5 | 5 | 1 | 5 | 3 | 5 | 7 | 0 | 4 | 18 | 6 | 26 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 10 | 4 | 0 | 1 | 4 | 0 | 8 | 1 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 6 | 0 | 2 | 6 | 0 | 1 | 4 | 1 | 7 | 5 | 0 | 1 | 5 | 4 | 12 | 4 | 6 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 3 | 0 | 2 | 6 | 1 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 3 | 8 | 1 | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 7 | 0 | 2 | 3 | 1 | 2 | 3 | 2 | 18 | 13 | 0 | 5 | 6 | 7 | 9 | 4 | 2 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 5 | 1 | 2 | 2 | 0 | 1 | 4 | 3 | 19 | 17 | 0 | 7 | 7 | 11 | 15 | 6 | 5 | 8
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 6 | 0 | 4 | 7 | 4 | 1 | 2 | 1 | 38 | 19 | 0 | 2 | 7 | 3 | 15 | 5 | 3 | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 3 | 0 | 2 | 4 | 1 | 0 | 0 | 0 | 3 | 4 | 0 | 1 | 2 | 1 | 6 | 0 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 4 | 10 | 0 | 6 | 5 | 3 | 0 | 2 | 2 | 38 | 18 | 1 | 9 | 21 | 12 | 18 | 2 | 8 | 7
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 11 | 0 | 7 | 10 | 3 | 0 | 3 | 5 | 30 | 16 | 0 | 3 | 17 | 20 | 22 | 6 | 8 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 1 | 3 | 3 | 2 | 1 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 3 | 1 | 0 | 1 | 5 | 3 | 6 | 0 | 2 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 7 | 3 | 1 | 2 | 4 | 4 | 6 | 1 | 1 | 2
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 3 | 0 | 8 | 6 | 0 | 2 | 7 | 11 | 9 | 1 | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 2 | 0 | 1 | 4 | 1 | 0 | 0 | 2 | 9 | 3 | 0 | 3 | 4 | 1 | 3 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 3 | 0 | 1 | 2 | 1 | 1 | 0 | 2 | 9 | 1 | 0 | 8 | 9 | 4 | 5 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 7 | 0 | 7 | 3 | 0 | 0 | 4 | 2 | 9 | 6 | 0 | 3 | 8 | 6 | 7 | 6 | 3 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 5 | 0 | 0 | 3 | 5 | 0 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 5 | 0 | 0 | 1 | 3 | 1 | 0 | 1 | 2 | 13 | 11 | 1 | 1 | 10 | 4 | 9 | 1 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 5 | 0 | 3 | 2 | 1 | 0 | 3 | 5 | 12 | 18 | 1 | 8 | 8 | 9 | 4 | 3 | 5 | 2
Dysaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 8 | 10 | 0 | 1 | 2 | 6 | 9 | 2 | 0 | 3
Freezing phenomenon (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 4 | 7 | 0 | 7 | 5 | 1 | 0 | 0 | 7 | 21 | 25 | 1 | 3 | 11 | 15 | 6 | 3 | 5 | 11
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 2 | 2 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 4 | 2 | 0 | 0 | 3 | 0 | 3 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mononeuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 3 | 0 | 1 | 2 | 0 | 1 | 1 | 2 | 4 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 2 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 6 | 3 | 0 | 0 | 3 | 2 | 4 | 2 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 3 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 1 | 0 | 8 | 7 | 5 | 4 | 1 | 3
Polyneuropathy (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3 | 1 | 1 | 1 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 2 | 0 | 1 | 4 | 1 | 1 | 2 | 2 | 11 | 8 | 0 | 4 | 7 | 3 | 4 | 2 | 2 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 6 | 10 | 0 | 0 | 1 | 1 | 2 | 2 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 4 | 1 | 2 | 3 | 1 | 0 | 1 | 3 | 6 | 7 | 0 | 3 | 4 | 3 | 9 | 1 | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 8 | 1 | 7 | 2 | 1 | 1 | 1 | 1 | 22 | 18 | 0 | 5 | 8 | 12 | 14 | 6 | 1 | 3
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 6 | 5 | 5 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 2 | 1 | 3 | 2 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 3 | 0 | 0 | 15 | 9 | 11 | 1 | 0 | 0
Micturition frequency decreased (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 5 | 0 | 1 | 3 | 4 | 1 | 1 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Breast haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nipple exudate bloody (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 2 | 1 | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 5 | 7 | 0 | 8 | 12 | 2 | 0 | 2 | 8 | 44 | 40 | 0 | 15 | 19 | 17 | 18 | 6 | 5 | 9
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 0 | 2 | 3 | 1 | 1 | 0 | 0 | 10 | 4 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 1 | 9 | 0 | 3 | 9 | 3 | 1 | 3 | 7 | 49 | 26 | 1 | 14 | 20 | 18 | 14 | 8 | 4 | 14
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 2 | 4 | 0 | 0 | 0 | 3 | 8 | 7 | 0 | 4 | 2 | 0 | 1 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 8 | 4 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 4 | 1 | 0 | 1 | 2 | 0 | 4 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 0 | 3 | 4 | 1 | 1 | 2 | 4 | 4 | 1 | 0 | 2 | 6 | 4 | 7 | 0 | 2 | 3
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 2 | 5 | 2 | 0 | 2 | 4 | 3 | 4 | 1 | 0 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 4 | 0 | 1 | 5 | 1 | 0 | 1 | 1 | 15 | 10 | 0 | 0 | 6 | 1 | 0 | 3 | 4 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 5 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 3 | 7 | 0 | 2 | 1 | 3 | 4 | 5 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 3 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 6 | 2 | 0 | 2 | 6 | 1 | 1 | 0 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 1
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 5 | 7 | 2 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 7 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 1 | 4 | 1 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 3 | 3 | 4 | 2 | 0 | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 8 | 1 | 2 | 0 | 0 | 3 | 0 | 1 | 1 | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 13 | 8 | 0 | 5 | 11 | 6 | 15 | 5 | 1 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 3 | 0 | 2 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 3 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 4 | 0 | 1 | 2 | 3 | 3 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 2 | 0 | 1 | 2 | 2 | 2 | 1 | 0 | 3 | 7 | 1 | 2 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1 | 4 | 13 | 0 | 13 | 16 | 2 | 1 | 7 | 11 | 34 | 43 | 1 | 8 | 28 | 32 | 34 | 17 | 12 | 9
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 6 | 5 | 1 | 10 | 9 | 2 | 0 | 3 | 12 | 15 | 25 | 0 | 7 | 6 | 15 | 13 | 3 | 5 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 3 | 1 | 8 | 6 | 2 | 0 | 1 | 4 | 12 | 23 | 0 | 5 | 19 | 15 | 22 | 13 | 3 | 6
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 1 | 1 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 2 | 2 | 1 | 3 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 6 | 3 | 0 | 2
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 1 | 5 | 1 | 3 | 3
Hypertension (Vascular disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 7 | 4 | 0 | 2 | 4 | 2 | 2 | 2 | 2 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 4 | 0 | 3 | 2 | 0 | 0 | 1 | 1 | 11 | 7 | 0 | 1 | 4 | 5 | 5 | 3 | 1 | 0
Lymphoedema (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 2
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-10-03): https://cdn.clinicaltrials.gov/large-docs/94/NCT01928394/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-12): https://cdn.clinicaltrials.gov/large-docs/94/NCT01928394/SAP_001.pdf